CLINICAL TRIAL: NCT00779688
Title: Endoscopic Retrograde CholangioPancreatography Endomicroscopy Registry Outcomes Database
Brief Title: A Registry of Patients Undergoing Cellvizio Endomicroscopy and Endoscopic Retrograde Cholangiopancreatography(ERCP) Imaging Procedures for Diagnosing Pancreatic and Bile Duct Cancers
Status: Completed | Type: Observational
Sponsor: Mauna Kea Technologies (Industry)
Collaborators: Cellvizio Inc. (Industry); Emissary International LLC (Industry)
Responsible Party: Anne Osdoit / Clinical Affairs Manager, Mauna Kea Technologies
Other Study IDs: MKT-2008-ERCP-01; WIRB 20081709
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Pancreatic Cancer; Bile Duct Cancer
Keywords: Endoscopic Retrograde Cholangiopancreatography; ERCP; bile duct cancer; pancreatic duct cancer; gall bladder; pancreas; duodenoscope; Cellvizio; endomicroscopy; cholangiopancreatoscopy; Biliary Tract Neoplasms (suspected); Biliary Tract Mass (suspected); Biliary Tract Stricture (suspected); Pancreatic Duct Neoplasms (suspected); Pancreatic Duct Mass (suspected); Pancreatic Duct Stricture (suspected)
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms; Biliary Tract Neoplasms | interventions — Microscopy, Confocal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Probe-based confocal laser endomicroscopy — ERCP with or without cholangiopancreatoscopy will be performed by the endoscopist as clinically indicated. If findings at ERCP and/or prior imaging studies and/or clinical assessment suggest possible malignancy and/or an indeterminate biliary or pancreatic pathology Cellvizio probe-based endomicroscopy will be performed during ERCP.
  Other Names: Cellvizio endomicroscopy; Confocal Laser Scanning Microscopy

SUMMARY:
This registry will collect data from patients routinely undergoing an ERCP and Cellvizio endomicroscopy procedure (and optionally an additional cholangiopancreatoscopy procedure) due to suspected pancreatic or bile duct cancer. The objective is to determine if endomicroscopy images collected using the marketed Cellvizio device may help endoscopists more accurately diagnose, in conjunction with traditional tissue sampling techniques, whether a suspected lesion is malignant or benign.

DETAILED DESCRIPTION:
This is a registry study to collect high quality longitudinal data from patients with suspected or indeterminate pancreaticobiliary pathology who are undergoing an ERCP with Cellvizio probe-based endomicroscopy procedure, with or without supplemental direct cholangiopancreatoscopy. The hypothesis is that ERCP with Cellvizio probe-based endomicroscopy improves differentiation of biliary and pancreatic duct lesions versus ERCP alone.

Direct measures of accuracy (sensitivity, specificity, etc.) in the differentiation of malignant versus benign biliary and/or pancreatic duct lesions will be compared for the combination of endomicroscopy and ERCP imaging and ERCP alone. These presumptive diagnoses will be compared against a 12-month follow-up confirmed histopathologic endpoint (an initially-benign pathologic diagnosis will be confirmed by a 12-month follow-up). Secondary objectives include collecting various safety and technical performance parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age
2. Willing and able to comply with Registry procedures and provide written informed consent to participate in the Registry
3. Indicated for ERCP and/or cholangiopancreatoscopy
4. Indeterminate or suspected biliary and/or pancreatic stricture, mass, or neoplasm

Exclusion Criteria:

1. Subjects for whom ERCP procedures are contraindicated
2. Known allergy to fluorescein dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Undergoing Cellvizio Endomicroscopy and Endoscopic Retrograde Cholangiopancreatography(ERCP) Imaging Procedures for Diagnosing Pancreatic and Bile Duct Cancers
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Comparative histopathology-confirmed measures of Cellvizio endomicroscopy and ERCP accuracy in the differential diagnosis of suspicious lesions. | 12-month diagnostic follow-up confirmation

CONTACTS AND LOCATIONS:
Overall Officials: Yang Chen, MD, FACP, FACG, Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (4):
  - University of Colorado Hospital, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Institut Paoli-Calmettes, Marseille, France
- Klinikum rechts der Isar, Munich, Bavaria, Germany